CLINICAL TRIAL: NCT02235376
Title: Criteria of Extubation Failure of Brain Injured Patients. Elaboration of a Prognostic Score.
Acronym: GODWEAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0201
Record Dates: First submitted 2014-07-28; First posted 2014-09-10 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Brain Injury
Keywords: Critical Care; Brain injured patients; Mechanical Ventilation; Weaning; Extubation; Prognostic score; Clinical examination
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- critical care
  Interventions: Other: weaning trial of mechanical ventilation

INTERVENTIONS:
Other: weaning trial of mechanical ventilation

SUMMARY:
Identification of criteria associated with extubation failure of brain injured patients. Elaboration of a prognostic score of extubation failure of brain injured patients.

DETAILED DESCRIPTION:
Prospective clinical study in ICU with brain injured ventilated patients eligible to extubation.

Identification of clinical and biological criteria associated with failure of extubation.

Elaboration of a prognostic score of extubation failure of brain injured patients, based on criteria previously identified with multivariate analysis.

Failure of extubation is defined by the need of re-intubation or the need for non-invasive ventilation within 48 hours or more after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Adult brain injured patients ventilated eligible to discontinuation of mechanical ventilation
* Stable respiratory and hemodynamic conditions
* Ventilated patients for more than 48 hours
* Adequate gaseous exchange (SpO2 ≥ 92% and respiratory rate ≤ 35/min, FiO2 ≤ 40%, positive end-expiratory pressure ≤ 5 cmH2O, pressure support ≤ 8 cmH2O, tidal volume ≥ 7mL/kg
* Therapeutic extubation

Exclusion Criteria:

* • Status epilepticus

  * Cerebrospinal infection
  * Patients under 15 years old
  * Mechanical ventilation of < 48 h
  * Spinal cord injury
  * Withdrawal of life support

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: brain injured patients
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Failure of extubation defined by the need of reintubation or the need for non-invasive ventilation | at day 2
  - Failure of extubation defined by the need of reintubation or the need for non-invasive ventilation within 48 hours or during ICU stay

SECONDARY OUTCOMES:
Severity scores (SAPS II, SOFA, GCS…) ) at patient admission in ICU | at ady 1
Cause of brain injury (traumatic, ischemic, hemorrhagic or post-operative) at patient admission in ICU | at day 1
Localisation of brain injury (hemispheric, supra- or sub-tentorial) at patient admission in ICU | at day 1
Complete neurological examination (Glasgow score, Coma Recovery Scale, FOUR score, cough, brain stem reflexes) just before extubation | at day 1
cardiologic history (cardiac insufficiency or ischemic cardiomyopathy) during ICU stay | at day 1
- Pulmonary examination (arterial gasometry, ventilatory parameters: mode, frequency, positive end expiratory pressure, inspiratory pressure, tidal volume, minute ventilation, oxygen level) just before extubation | at day 1
- Cause of extubation failure before 48 hours (respiratory, hemodynamic, aspiration, ...) | at day 2
Delay of extubation from intubation day (number of days) | at day 1
Glasgow Outcome Score (GOS) | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell CHABANNE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France